CLINICAL TRIAL: NCT03687294
Title: Diagnostic Accuracy of Human Transcriptional Activator(MYB) Expression by ELISA Technique Versus Immmunohistochemistry in Detecting Salivary Gland Carcinomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yousra Refaey, pricipal investegator, Cairo University
Other Study IDs: yousrarefaey11
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Malignant Neoplasm of Salivary Gland; Benign Neoplasm of Salivary Gland
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group I: patients suffering from malignant salivary gland tumors.
  Interventions: Device: enzyme linked immunosorbent assay (ELISA)
- Group II: patients suffering from benign salivary gland tumors.
  Interventions: Device: enzyme linked immunosorbent assay (ELISA)

INTERVENTIONS:
Device: enzyme linked immunosorbent assay (ELISA) — ELISA measure MYB in tissue biopsy in benign and malignant salivary gland tumors

SUMMARY:
in this resarch we will use ELISA Technique to estimate Human Transcriptional Activator(MYB) Expression .compare it by Immmunohistochemistry analysis of MYB Expression in the malignant and benign salivary gland tumor

ELIGIBILITY:
Inclusion Criteria: .

* Patients with clinically evident salivary gland tumors; malignant tumors will be recruited in group I
* Benign tumors will be recruited in group II.

Exclusion Criteria:

* Subjects taking any drugs inducing any changes that could affect the salivary glands.
* Pregnant females.
* Subjects having any allergies, infectious or autoimmune diseases.
* Subjects having any metabolic disorders that can be manifested with salivary gland swelling as diabetes mellitus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian population
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-01-12 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Human Transcriptional Activator(MYB) Expression by ELISA Technique Versus Immmunohistochemistry in Detecting Salivary Gland Carcinomas | two years
  Diagnostic Accuracy of Human Transcriptional Activator(MYB) Expression by ELISA Technique Versus Immmunohistochemistry in Detecting Salivary Gland Carcinomas.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No